# Effect of early rehabilitation using an active/passive cycling device on muscle wasting in the critically ill:

## A randomised controlled pilot study

## Short Title - Muscle Wasting in the Critically III.

Turton P, Dyson S, Jenions L, Barrett-Jolley R, Gunther M, Connolly B,
Welters ID

Dr Peter Turton, MBChB(Hons) MPhil FRCA

Version 19.0, 15th June, 2018 (FINAL)

IRAS Number: 235656

## 1. Signature page

| Professor I. Welters, Chief Investigator |
|------------------------------------------|
| Dr P Turton, Academic Clinical Fellow |
| Karen Williams, Lead Research Nurse |
| Other selection |

Other staff:

Please see delegation log

| Name | Role | Signature |
|------|------|-----------|

| ICU-Acquired Weakness<br>15 <sup>th</sup> June 2018 | Study Protocol – Version 19 | P. Turton, I. Welters |
|---|---|---|
| Contents | | |
| Title page | 1 | |
| Signatures | 2 | |
| Contents | 3-4 | |
| Abbreviations and definitions | | 5-6 |
| Summary | | 7-8 |
| Background | | 9-14 |
| ICU Acquired Weakne | ess | 9-10 |
| Physical methods of p | reventing and treating muscle loss | 9-12 |
| Scientific rational | 12-14 | |
| Trial objectives and purpose | | 15-20 |
| Research questions | 15-17 | |
| Study design | | 17 |
| Subject selection | | 17-19 |
| Subject recruitment | | 19-20 |
| Trial interventions and invest | igations | 21-25 |
| Patient end points | 25 | |
| Data to be collected | 25 | |
| Other data collected | 27 | |
| Further laboratory studies | 28 | |
| 3 Page | | |

| ICU-Acquired Weakness<br>15 <sup>th</sup> June 2018 | Study Protocol – Version 19 | P. Turton, I. Welters |
|---|---|---|
| Statistical analysis | | 28-29 |
| Blinding | | 29 |
| Ethical considerations | | 29-30 |
| End of study, disseminate | 30-31 | |
| Appendix A – Study flow | diagrams | 32-33 |
| Appendix B – The CYCL | E trial exclusion criteria | 34-35 |
| Appendix C – Proposed | measurements and statistical tests | 36 – 38 |
| References | | 39-43 |

#### Abbreviations and definitions

6MWT Six minute walk test

APACHE II Acute Physiology And Chronic Health Evaluation II

BMI Body Mass Index

CAM-ICU Confusion Assessment Method for the ICU

DTF Diaphragmatic Thickening Fraction (the ratio of muscle

thickness at expiration compared to inspiration).

FES Functional Electrical Stimulation

FEV<sub>1</sub> Forced Expiratory Volume in 1 Second

FVC Forced Vital Capacity

Hz Hertz – a unit of frequency required for FES

ICNARC Intensive Care National Audit & Research Centre

ICU Intensive Care Unit

ICU-AW Intensive Care Unit Acquired Weakness

IL (6, 8, etc) Interleukin

mA Milli-amperes – a unit of current required for FES

MRC Medical Research Council. In this context it refers to the MRC

Sum Power Score, a subjective scale testing power in major

muscle groups.

NMES Neuro-muscular Electrical Stimulation

| <b>ICU-Acquired Weakness</b> |
|------------------------------|
| 15 <sup>th</sup> June 2018 |

Study Protocol – Version 19

P. Turton, I. Welters

PFT Pulmonary Function Test

SF-36 Short Form Health Survey (with 36 items)

SOFA Sequential Organ Failure Assessment

## Summary

The aim of this randomised controlled pilot trial is to assess whether a 14-day course of cycling with Functional Electrical Stimulation (FES) can prevent muscle loss and preserve muscular function in septic patients who are sedated, intubated and mechanically ventilated in the ICU, compared to a control group of patients who will receive standard daily physiotherapy.

It is known from several studies that muscle size significantly decreases early in a patient's admission to critical care with sepsis. This rapid muscle loss is likely due to a combination of disuse atrophy and systemic inflammation. Passive movement and stretching exercises performed by physiotherapists, do not appear to prevent muscle loss. Previous studies with electrical nerve stimulation have provided mixed results with respect to preserving muscle thickness. The proposed study differs from previous investigations in that we will use a cycling device which passively moves the participants legs whilst they are in bed, sedated and on a breathing machine, but with the addition of low current electrical stimulation applied on leg muscles, so that they can contract and relax in time with the movement of the cycle, thus providing "functional stimulation" rather than just electrical stimulation.

Briefly, we intend to enrol participants into the study within 48 hours of being intubated and mechanically ventilated for sepsis. Ultrasound measurements of the leg muscles, abdominal musculature and diaphragm will be performed, alongside baseline blood and urine sampling. Muscle biopsies will be taken from the leg before and after the 14-day study period. These biological samples will serve to investigate cellular mechanisms involved in muscle wasting as part of a separate translational follow-up research project.

This pilot study includes ultrasound measurements of different muscle groups and clinical outcomes in the intervention and control group and will allow us to define the most pragmatic and clinically relevant primary outcome measure for larger multicentre trials.

Those randomised to the intervention will be in the study for 14 days. They will receive five 30 minute treatments with the device per week. Therefore in a 14 day period, they should receive 10 treatments.

Repeat ultrasound measurements will be taken on days 3, 5, 7, 10 and 14. Further blood and urine samples will be taken on days 5, 10 and 14. A second muscle biopsy will be taken on day 14.

Should patients be liberated of mechanical ventilation before day 14, they will continue in the trial, providing that they provide consent to do so.

All survivors from the trial will be invited to a follow up study 3 months from hospital discharge, where further ultrasound assessments, plus assessment of balance, strength and psychological wellbeing will be assessed.

There are two broad aims to this study. The first is to identify the clinically most useful measurement of changes in muscle size by investigating a number of muscle groups, using several indices of muscle size. This will inform us of the most suitable primary outcome for further follow-up studies.

The second aim is to assess the safety profile and feasibility of the study.

Specifically, we will determine the number of successfully completed cycling

sessions, identify logistical hurdles and patient safety risks, such as haemodynamic deterioration or accidental extubation.

## **Background**

## **ICU Acquired Weakness**

Intensive Care Unit Acquired Weakness (ICU-AW) is a common and potentially debilitating consequence of admission to an intensive care unit with critical illness(1). It is defined as a diffuse generalised muscle weakness without a readily identifiable cause, which occurs after developing a critical illness. Nerve conduction studies and electromyography often demonstrate both polyneuropathy and myelopathy(2). Patients with critical illness, having survived the initial acute insult, are often left with long term problems with mobility(3), which preclude independent living even five years after hospital discharge(4). These long-term sequelae represent a massive burden on both the health service and the patients' families and caregivers in the community(5).

Muscle size, expressed as either muscle thickness or muscle cross-sectional area of muscle in the limbs, can be easily tracked using bedside ultrasound methods(6). As well as size and cross-sectional area of muscles, further information, such as the arrangement of fascicles within the muscle (known as the muscle architecture)(7) and ultrasound echogenicity(8), can also be easily obtained at the bedside. Echogenicity is helpful in determining infiltration of muscle with fat or fibrosis, which usually occurs as a result of disease or aging(9). These methods have been shown to have good reliability and accuracy in adult critically ill patients(10). Our own work has demonstrated that patients lose over 10% of their muscle thickness in the first 96 hours of mechanical ventilation, and that by 10 days, 28% of muscle thickness was lost(7). Changes to the arrangement of the fascicles within the muscle also occur, with pennation angle reducing over time, suggesting that weakness may occur

through loss of force generation as a result of smaller pennation angles. These results are in keeping with another recent study which demonstrated a 30% reduction in muscle thickness in the vastus intermedius in critically ill patients over 10 days(6) and far exceeds the previously demonstrated loss of 8% muscle thickness over five weeks bed rest in healthy volunteers(11). Ultrasound measurement of the quadriceps femoris muscle has shown a negative relationship between length of stay in critical care and muscle size during the admission(12). These structural changes are associated with loss of individual fibre area, increased loss of protein, and decreased protein synthesis, in comparison to healthy controls(13).

## Physical methods of preventing and treating muscle loss

## Supine cycling

Early mobilisation of patients has been shown to improve to outcomes in patients who survive critical illness(14). There are randomised control trials being carried out at present, looking at supine cycling in patients in critical care(15). Such cycling sessions can be active (entirely initiated by the patient), passive (the patient's legs are moved for them by the cycle, but no effort comes from the patient,) or assisted (where the patient makes the initial effort to move, and is then supported by the cycling device). Previously reported smaller trials have shown that the technique is safe, can be carried out in sedated patients, and can be performed safely whilst the patient is receiving intravenous infusion therapies(16). Another randomised control trial, the MoVe-ICU study, is currently in progress, examining how passive cycling in the early stages of critical illness will change the muscle morphology and ultrasound

appearance of leg muscle in these patients(17). It is, however, currently known whether early passive cycling during critical illness compared to standard treatment does improve 6-minute walk test scores in patients who survive critical illness(18).

## **Neuromuscular stimulation**

Neuromuscular electrical stimulation (NMES) has been shown to improve muscle strength and balance in patients outside of ICU, for example stroke survivors(19). NMES used in patients after discharge from ICU resulted in no difference in muscle layer thickness, but did recover muscle strength more quickly compared to controls(20). In patients who received NMES whilst still mechanically ventilated, walking distance on discharge was greater than those receiving a sham therapy, but there was no difference in lower limb extremity muscle strength(21). The technique itself however has been shown to be safe and simple to carry out(22).

#### **Functional Electrical Stimulation**

Functional electrical stimulation (FES) also involves the use of electrically stimulating the muscles of the leg, but has been combined with a cycling device in order to carry out supine cycling exercises in patients who are still sedated. This device has been trialled in stroke patients, where it has improved muscle strength and function outcomes in a number of settings(23)(24), in comparison to passive cycling. Gait and posture have also been shown to improve after FES cycling(25).

In the critical care population, a case-control study has shown that FES with cycling improves physical function and reduces the incidence of delirium(26).

15<sup>th</sup> June 2018

NMES and FES, whilst both using electrical current to stimulate muscle contraction, are distinct treatment modalities. NMES requires the delivery of low voltage electricity to muscles directly underneath surface electrodes which are placed on the skin(27). Studies using NMES have focussed on one muscle group per study. FES differs from NMES in that different muscle groups are stimulated in an alternating pattern. The addition of cycling allows for a muscle group to be recruited via electrical stimulation, whilst its antagonistic muscle group is relaxed. This stimulating pattern is then reversed so that the relaxed muscle is contracted, and the contracted muscle is relaxed.

There is an on-going randomised control trial, (eStimCycle – Early Rehabilitation in Critical Care, register with clinicaltrials.gov, trial identifier NCT02214823) in which patients with sepsis who are mechanically ventilated for longer than 48 hours, are being randomised to receive FES with cycling in one leg, with the other leg receiving no FES but still undergoing passive cycling, or randomised to a control group of standard physiotherapy(28). Our proposed trial will differ in the following ways:

- Both legs will be treated with FES with cycling. Comparison will be made with a separate control group receiving standard physiotherapy.
- In addition, the rectus abdominis muscle will be stimulated to assess if core muscle strength improves.
- The effects on other organ systems, including changes to the diaphragm and anterior abdominal wall muscles, will be investigated alongside changes to the lower limb. These are detailed in the methods section.

#### Scientific rationale

Immobility, independently of illness, leads to rapid muscle wasting. This atrophy is largely mediated through transcription of a range of "atrogenes"; including elements of the autophagic and ubiquitin proteasome systems(29). The final common path appears to be similar in disuse in volunteers and in ICU-AW patients, but in disease states additional intracellular pathways lead to atrogene transcription, resulting in a more rapid and exaggerated atrophy. Direct comparison of immobilised or bedrested healthy individuals with ICU-AW patients are plagued with numerous confounding variables, but as a guide the former may lose 0.6% muscle size per day, whilst our data show that ICU-AW patients routinely loose about 2.5% per day(7). This figure is similar to the loss of force seen (thumb muscle) in ventilated critical care patients (30% over 14 days)(30).

In healthy individuals exercise promotes synthesis of muscle contractile proteins and supresses a range of pathways that induce atrogene transcription. In a wide range of diseases, cytokines activate the NFkB system that in turn promotes atrogenesis. The role of NFkB signalling itself is complex with both exercise and disuse reported to increase activity(31)(32)(33)(34)(35). Reactive oxygen species (ROS) are elevated in older, frail people, and this also triggers NFkB activation(36). A further pathway leading to atrogene transcription is myostatin-SMAD. This system is activated in a number of situations including ageing and critical care, but its physiological regulation is largely unknown(37). Therefore, a typical older ICU-AW patient will have a conflagration of several different intracellular pathways that lead to autophagy, mitochondrial and myofibril degradation. In this project, we will use muscle biopsies from patients undergoing FES with supine cycling, and control patients to identify the intracellular pathway changes that underlie muscle

preservation. In particular, it is important that we identify which intracellular pathway changes correlate with muscle preservation, or lack thereof, so that future intervention studies can establish whether this relationship is causal and devise novel therapeutic interventions that could be deployed independently of FES.

Cytokines have been implicated in the development of ICU-AW, and a recent study has shown that in a cohort of patients who developed ICU-AW, high levels of the interleukin (IL) -6, IL-8, IL-10 and fractalkane were found, in comparison to critically ill patients who did not develop ICU-AW(38). Raised cytokine levels may cause muscle damage through poor oxygenation of muscle(39). This may potentially be explored via a non-invasive infra-red spectroscopy technique(40).

## Trial objectives and purpose

The main objective is to perform a randomised controlled pilot study to assess the effects of daily cycling with functional electrical stimulation in sedated and mechanical ventilated intensive care patients. We will measure several indices of muscle size in a number of muscles groups over a 14-day period. The second objective is to assess the feasibility of the study protocol, so that if required, study procedures can be refined for a definite randomised control trial.

Justification for a pilot study:

A wide variation in the use of electrical stimulation in the critically ill and the effects on muscle thickness has been reported in previous studies. A structured review found four studies, each assessing the effect of electrical stimulation on different muscle groups(41). Whilst two studies found that the muscle studied decreased, even with stimulation, a third study found no change to the size of the muscle, whilst a fourth demonstrated and increase in size. Furthermore, a study of critically ill patients on muscle wasting in the abdominal muscles, demonstrated that electrical stimulation slowed muscle loss in the critically ill compared to patients who did not receive it(42). The potential to increase thickness of abdominal muscle groups with neuromuscular stimulation has been demonstrated before, albeit in healthy volunteers(43). A pilot study, consisting of a number of muscle groups and measurement parameters, would allow us to refine the protocol to define the most pragmatic and clinically relevant primary outcome measure for a later definitive trial.

## Research objectives:

Research objectives regarding muscle thickness and function:

- 1. What is the effect of a 14day course of 30 minutes cycling with functional electrical stimulation, consisting of 10 treatments over 14 days, on muscle thickness, cross-sectional area, fascicle pennation angle, fascicle length and echogenicity of the following muscles, compared to a control group receiving standard daily physiotherapy:
  - a) Vastus lateralis all measurements
  - Rectus femoris, vastus medialis, vastus intermedius cross sectional area and echogenicity
  - c) Medial head of gastrocnemius all measurements
  - d) Rectus abdominis Cross section area and echogenicity
  - e) Diaphragm muscle thickness, thickening fraction and maximal excursion
- 2. Are such differences between treatment and control group maintained 3 months after hospital discharge?
- 3. Does treatment with FES and cycling affect other organ systems, as defined by requirement for renal replacement therapy, inotropic/vasopressor support, time to wean from ventilation, and incidence of delirium?
- 4. Do ultrasonic muscle changes correlate with biochemical alterations measured in serum and muscle tissue? The details of these changes will be described in a separate study protocol.

Research objectives to assess feasibility and patient safety:

- How many of the 10 sessions can be successfully completed in a 14-day period? Successful completion will comprise at least 20 min of cycling activity.
- 2. What are the reasons for missed or incomplete treatment sessions?
- 3. What is the incidence of adverse effect such as haemodynamic changes (blood pressure or heart rate) of more than 20% baseline, central or arterial line dislodgement, accidental extubation or falls?

## Study design

We intend to perform a randomised control pilot trial with two arms: 1. Patients receiving standard physiotherapy will serve as a control group, 2. Patients undergoing FES plus supine cycling 5 times per week. In a number of muscle groups, muscle thickness will be measured with ultrasound to determine the clinically most useful index to describe changes in muscle size during treatment with 10 sessions of FES with cycling over a 14-day period.

## **Subject selection**

Patients will be recruited in the Intensive Care Unit of the Royal Liverpool University
Hospital. All patients will be over 18, and have a critical illness that requires
mechanical ventilation with an initial period of sedation. This study will focus on
patients with a definite or suspected case of sepsis from any source.

Sepsis has been recently redefined as: "Life threatening organ-dysfunction caused by dysregulated host response to infection" whilst septic shock has become a subset

of sepsis, defined as: "circulatory and cellular/metabolic dysfunction associated with a higher risk of mortality(44).

For the purposes of this study, a patient will be regarded as septic if they have evidence of infection-related organ failure (e.g. sepsis-associated coagulopathy, altered mental state, cardiovascular dysfunction, acute kidney injury, and altered liver function) and require invasive mechanical ventilation with either definite or suspected evidence of infection. This is to allow prompt treatment with FES rather than waiting for a positive microbiological result to be obtained.

Within the definition of sepsis "from any source" a list of following is illustrative but not exhaustive:

- Urogenital sepsis (including urosepsis, pyelonephritis, endometritis and chorioamnionitits)
- Pneumonia (including community acquired, hospital acquired, and aspiration pneumonia. Ventilator associated pneumonia would be excluded.)
- Neurological infections such as encephalitis and meningitis.
- Cellulitis, osteomyelitis and infections of soft tissue NOT affecting the lower limb.
- Surgical infections, including post-operative laparotomy with evidence of peritoneal soiling, and evidence of infection prior to the operation, in patients who require 2 or more organ system support after the operation.
- Intra-abdominal sepsis, including biliary sepsis, hepatitis, and acute
  pancreatitis. In the case of acute pancreatitis, evidence of infection is
  required to fulfil the criteria. Acute pancreatitis with sterile tissue/fluid samples
  would not be suitable.

#### Exclusion criteria include:

- Patients under 18
- Patients who decline consent
- Pregnancy
- Neuromuscular disease
- Rhabdomyolysis
- Lower limb trauma
- Patients unlikely to survive to 96 hours post admission
- Consent unobtainable within 48 hours of admission
- Morbid obesity (BMI>40).
- Presence of a pacemaker or Implantable Cardiac Defibrillator (ICD).
- Unlikely to be mechanically ventilated for more than 48 hours.

## Subject recruitment

Patients will be mechanically ventilated and sedated and therefore unable to consent to the trial. The patient's next of kin will be approached to act as a consultee, to provide consent for the patient to take part in the study. If the patient regains capacity to consent for themselves, they will be informed about their participation in the study and retrospective consent will be sought.

The process for taking consent from the next of kin is as follows:

Patients will be screened every morning by the research nursing team to identify potential patients who meet the inclusion criteria. Eligible patients will be discussed with the medical team that day to assess if the medical condition or comorbidities

preclude recruitment into the trial (for example, the medical team have decided to withdraw care).

The next of kin will be approached by a member of the research team. The aims of the study and a discussion of what would happen to their relative during the trial will take place, and an information leaflet will be given to the next of kin. At this point, there is no obligation to sign a consultee declaration form. The next of kin will be given time to think about whether they want their relative to take part, and they can discuss the study with other members of the family.

Once the next of kin has decided to provide consent, they will sign a consultee declaration form, acting as a consultee on behalf of their relative. Should they later decide to withdraw this declaration, the patient will be withdrawn from the study, and all samples and data will be disposed of.

Once the patient regains capacity, they will be approached by the research team, explaining the involvement in the study so far, the aims of the study, and what will happen if they agree to continue in the study. They will again be given time to think about whether they want to continue in the study, and will be given an information leaflet to read. There is no time limit on this, and once ready, the patient will have to provide retrospective consent by signing the appropriate retrospective consent form. Should they decide they do not want to take part in the study, all further cycling sessions would be cancelled. An added option has been incorporated into this form, in the event that the patient decides they do not want any more cycling sessions, but that we can continue to store and use blood, urine and muscle biopsy samples, and that no further samples will be taken. In the event that they do not consent to us using pre-existing samples, and they do not want any further cycling sessions, then

all samples will be destroyed. This includes the deletion of ultrasound images from any storage medium.

Where a next of kin cannot be contacted within 36 hours of admission, a professional consultee declaration by the patient's clinical team will be considered to allow recruitment into the study within the 48h time frame. The senior clinician in the medical team will be provided with an information leaflet, and when ready, will be given a Nominated Professional Consultee Declaration form to sign.

Patients for whom a consultee declaration form cannot be signed within 48h after intubation, will need to be excluded from the trial.

## Trial interventions and investigations

The day on which a valid consultee declaration is obtained, will be classified as Day 0. Within 24 hours, patients will receive an ultrasound of the vastus lateralis to assess muscle thickness and fascicle pennation angle, and ultrasounds of the four heads of the quadriceps (rectus femoris, vastus lateralis, medialis and intermedius), medial head of gastrocnemius, rectus abdominis and diaphragm. Blood and urine samples will be taken from pre-existing arterial (or central venous) lines and urinary catheters. A percutaneous muscle biopsy will also be taken under sedation and local anaesthesia from the vastus lateralis muscle. All samples will be obtained on study day 1 before the intervention is started.

Ultrasound scanswill be repeated on days 3,5, 7, 10 and 14. Our work and previous publications suggest that significant losses in muscle thickness can be detected by

ultrasound as early as day 5, and are more pronounced by day 10. Further blood and urine samples will be taken on days 5, 10 and 14.

Ultrasound scanning of the following muscles will take place on day 1:

- Vastus lateralis
- Rectus femoris Vastus lateralis, intermedius and medialis (cross section area).
- Medial head of gastrocnemius
- Diaphragm
- Rectus abdominus

All ultrasound scans will be taken with the patient lying supine. Vastus lateralis and rectus femoris imaging will be performed with the limbs straight and in contact with the bed. Gastrocnemius scans will be taken with hip and knee flexed so that the foot is in contact flat with the bed. These methods have been used in our previous study(7) and have been cited in other work(45). Diaphragmatic ultrasound will include diaphragmatic thickness, Diaphragmatic Thickening Fraction (DTF) and diaphragmatic excursion on both sides according to standard procedures.

Muscle biopsies will be taken percutaneously under local anaesthetic, on days 1 and 14 only.

After the initial samples have been taken, the patient will be randomised using a computer-generated randomisation system, to receive either FES plus cycling or standard physiotherapy. A computer-based block randomization system will be generated using R (randomizeR: An R Package for the Assessment and Implementation of Randomization in Clinical Trials). Allocation concealment will be

guaranteed by management of the randomization table by an external company not involved in the conduct of the study (MoRe Data GmbH, Giessen, Germany). Patients receiving FES plus cycling will receive 30 minutes of FES cycling on 5 days per week. Other studies have applied between 20 -50 minutes of this exercise. The device to be used is the Restorative Therapies (RT) 300 Supine with FES system, plus a 12 channel SAGE stimulator (Restorative Therapies Ltd, Baltimore, Maryland, USA). Surface electrodes will be placed on the quadriceps, hamstrings and calf muscles of both legs, with an additional electrode placed across the rectus abdominis muscle. The aim of the electrical stimulation is to produce visible contractions in each muscle group, without causing pain. If a contraction cannot be seen, treatment will continue, but with regular palpation of the muscle groups to feel for contraction. This will be done every 5 minutes throughout the intervention period. In line with eStimCycle study, a maximum current of 140mA, pulse duration of 250-500 microseconds, frequency of 40 Hz and pedal cadence of 30-45 revolutions per minute will applied. The intervention will be performed within 24h after consent has been obtained and will be classified as study day 1. Study day 1 has to occur within 72 hours of intubation. Patients will receive the intervention on 5 days per week. There will be one cycling device on the Intensive care Unit, which can be used for 6-8 cycling sessions per day. Hence a total of up to 16 patients can be included at any given time point (6-8 patients in the interventional arm, 6-8 patients in the control group).

Patients will be fully monitored during the study, with standard ICU equipment, including electrocardiogram, heart rate, arterial blood pressure, end-tidal carbon dioxide tension and haemoglobin oxygen saturation. Heart rate variability will also

be measured using a skin sensor device (Isansys Lifecare Ltd, Abingdon, Oxfordshire, UK).

All patients randomised to the intervention arm will have cycling sessions with FES for 14 days. They will receive 5 sessions per week, and so should receive 10 sessions over a two week period. Should the patient be liberated from mechanical ventilation, they will carry on receiving cycling with FES until day 14. In the unlikely event that they cannot tolerate FES once extubated, the intervention will be stopped. Based on discussions with the manufacturer, we expect that less than 10% of patients would be unable to tolerate FES whilst extubated, however, we wish to confirm this statement as part of this pilot trial to inform future studies..

All patients, regardless of intubation status, will have no further sessions of FES after day 14. No further ultrasound scans, blood or urine tests will be conducted after day 14.

Ultrasound scans performed on day 14 will serve as the main comparator to baseline investigation.. In patients who failed to tolerate the intervention, ultrasound measurements will give an opportunity to assess if muscle is lost whilst not receiving FES, but still critically ill.

Patients with a tracheostomy allocated to intervention will also receive FES with cycling until day 14.

On day 14, in patients that are awake and suitably co-operative, assessment of strength using both hand grip dynamometry and the MRC Sum power score will be conducted by blinded physiotherapists.

Follow up testing will occur at 3 months post hospital discharge. This will include:

- Ultrasound of the 4 heads of the quadriceps and gastrocnemius muscles.
- Ultrasound of the diaphragm muscles.
- Performance of balance and gait testing using an electronic pressure detecting plate.
- Performance of a 6-minute walk test.
- MRC sum power test
- Handgrip strength using portable dynamometry
- Assessment of quality of life, using the SF-36 scale The SF-36 questionnaire is commonly used for follow-up in research studies involving critically ill patients and is routinely used in our follow-up clinics, to which patients are invited to attend 3 months after ITU discharge. If patients are not available to attend the follow-up clinics, an attempt will be made to obtain the SF-36 information via telephone interview. Patients will have the opportunity to decline participation.

There will be no procedure for breaking the codes for randomisation, as the study team and the patient cannot be blinded to the treatment allocation.

## **Patient end-points**

A patient will be removed from the study if:

- A relative withdraws consent on behalf of the participant.
- The patient, after regaining capacity, withdraws consent.

There is difficulty in complying with treatment with more than two treatment sessions per week being missed (e.g. due to haemodynamic instability).
 Criteria for a patient to not receive a cycling session are in line with the CYCLE trial<sup>15</sup>.

## Data to be collected

- Muscle cross sectional area, muscle thickness, muscle fascicle length,
   pennation angle and echogenicity in the vastus lateralis and medial head of
   gastrocnemius, change in muscle thickness and echogenicity of the rectus
   abdominus, diaphragm and change in cross sectional area of the rectus
   femoris and the three vastus muscles. These will be measured on days, 1, 3,
   5, 7, 10, and 14.
- Relationship between changes in muscle thickness and expression of blood and muscle inflammatory markers.
- Measures of balance and posture using a specialised balance board in patients who survive to discharge from ICU. This will be tested 3 months after hospital discharge.
- Long term outcome measures, including ultrasound measurement of ALL
  muscle groups, and tests of balances and gait, re-testing of the MRC Sum
  Power Score, and 6-minute walk test. Quality of life assessment will be
  conducted using the SF36 questionnaire.
- Ultrasonographic changes in diaphragmatic thickness, DFT and diaphragmatic excursion
- Incidence of delirium, as assessed by the CAM-ICU method.

 Data collected from routine monitoring, such as heart rate, heart rate variability, haemoglobin oxygen saturation and end tidal carbon dioxide tension.

#### Other data collected

To answer the secondary research questions, the following data will also be collected:

- Age, sex, weight, height, and Body Mass Index (BMI)
- Admission APACHE II, ICNARC and SOFA scores
- Routine blood results, including full blood count, urea and electrolytes, liver function tests, clotting screen and arterial blood gases.
- A daily diary of standard physiotherapy received, time taken, and treatment received.
- A daily diary of FES and cycling, including time spent cycling.
- Blood glucose measurements.
- Total infusion volumes, including inotropes/vasopressors, insulin, sedative agents, intravenous fluids, nasogastric feed and total parenteral nutrition.
- Documented evidence of delirium, as assessed by the CAM-ICU method.
- Ventilator settings, including inspired oxygen concentration, and time to wean off mechanical ventilation.
- Use of renal replacement therapy, mode of replacement and indication for replacement.
- Microbiological samples for culture.

- A "safety log" of incidents and injuries sustained in the course of using FES with cycling.
  - Dislodgement of arterial lines, central lines, urinary catheter and endotracheal tubes.
  - Haemodynamic changes including changes in blood pressure or heart rate of more than 20% of baseline.
  - o Falls
  - Other injury to staff or patients
  - Death
- Dose of cardiovascularly active drugs (inotropes, anti-arrhythmics, vasopessors)

## **Further laboratory studies**

As well as expression of cytokines and histones in both blood and muscle samples, muscle biopsies will be used to conduct single fibre contractility studies. Using the blood and muscle cytokine and histone levels, we can assess if contractility in these fibres is reduced in patients who have greater levels of inflammatory markers. Haematoxylin and eosin (H&E) staining will also be performed, to assess nuclei count, extra-cellular matrix production and muscle area.

Blood samples will be analysed by ELISA for a panel of cytokines (including muscle specific cytokines, 'myokines') and biopsies will be subject to RNA-sequencing to allow analysis of genome differentially transcribed genes independently of bias. Key members of differentially expressed gene pathways will be verified by qPCR and Western blots. To investigate whether differentially expressed genes result from

change in cytokine abundance, we will simulate this system *in vitro*. Cultured human muscle cells will be exposed to the observed differentially expressed cytokines and RNA-sequenced.

All laboratory investigations on samples obtained in this trial are part of a different funding and research application.

## Statistical analysis

In general, sample size calculations are not required for pilot studies. We chose to continue recruitment until 18 patients in each group have reached day 14 of the study. This design will allow us to calculate a realistic drop-out rate for future trials and thus assess feasibility. We will use the inclusion/exclusion criteria we anticipate using in follow-up trials. With 18 patients in each arm completing the study until day 14, we anticipate that useful information about the feasibility, the safety and the changes in muscle thickness can be obtained.

Although not the primary aim of this project, the results from this pilot study may be used to generate data for sample size calculations for larger follow-up trials.

Our previous non-interventional study showed a 50% drop out between days 1 and 10. Therefore, we anticipate recruitment of 36 patients per arm to achieve completion of the trial until day 14 in 18 patients.

The following estimates were considered for drop-out: Loss of 14-day follow-up due to death (10%), discharge from Intensive Care or High-Dependency Units before day 10 (10%), inability to tolerate the intervention (20%), decline to continue in the trial after regaining capacity (10%).

A detailed breakdown of all measurements preformed at different time points and the proposed statistical approach is listed in Appendix C.

In all statistical analyses, a p-value of less than 0.05 will be considered statistically significant. For multiple testing the Bonferroni-Holm correction will be applied.

## **Blinding**

Due to the nature of the study, it is not possible to blind the participants or the investigators. However, ultrasound images will be saved as numbered images, with no detail as to which group the images come from. Measurement of muscle thickness will be measured on a computer rather than at the bedside with ultrasound machine, so that the measurements are performed blinded.

## 2.2.9 Ethical considerations

Considerations related to subject selection and recruitment have been described already.

Blood samples and urine samples shall be taken from the patients indwelling arterial/central lines and urinary catheters. Surplus blood samples from blood taken for routine clinical purposes will be collected daily from the Clinical Chemistry Department. Should an arterial line or central line be unavailable, blood will be obtained from venepuncture, if possible as part of a daily routine venepuncture to minimise pain and infection risk. Urine sampling will be performed via an indwelling urinary catheter or via collection a urine sample at the bedside.

Muscle biopsies taken percutaneously may cause pain, skin infection, muscle and fat infection and bleeding. The risk of skin infection in one trial is 1in 800(46), and serious bleeding reported in 1 in 5000 cases(47).

## End of study, dissemination and archiving

The study is expected to start on August 1<sup>st</sup>, 2018. The study is expected to run for 2.5 years, ending on the 1<sup>st</sup> February 2021. The recruitment period is expected to last 12-18 months with expected recruitment of 2 patients/week. Data analys and final report will take 6 months. The suggested study period will allow a 3 month follow up appointment, within the 2.5 years. An interim analysis will take place after 50 patients will have been recruited.

The study will be ended early in the event that:

- Inability to recruit patients within 3 months after opening the trial.
- Serious adverse effects associated with the trial device
- Decision of the Data management committee after interim analysis
- The study sample is completed

Data will be presented at local, national and international conferences, as well as for publication in journals. Patients who took part in the study can have their results discussed at the 3 months follow up appointment, and will also be sent copies of any publication on request.

After data analysis is completed, all study material will be archived using an approved archiving company, in this instance Manchester Retrievals.

## Appendix A - Study Flow Diagram

## Recruitment, randomisation and groups



## Notes:

Patients may be extubated between day 1 and 14. If they are, they will continue to receive FES with cycling whilst awake. In the unlikely event that they cannot tolerate this, they will receive passive cycling without electrical stimulation until day 14.

Even if a patient is still intubated by day 14, the intervention will stop at day 14.

Follow up testing will occur at 3 months post hospital discharge.

## Time scale of investigations and interventions

| Procedure/Test | Day | Day | Day | Day | Day | Day | Day 14 | F/U |
|----------------|-----|-----|-----|-----|-----|-----|--------|------|
| | 0 | 1 | 3 | 5. | 7 | 10. | | 3/12 |
| Consent | х | | | | | | | |
| Randomisation | | X | | | | | | |
| Start | | X | | | | | | |
| Intervention | | | | | | | | |
| Urine | | X | | X | | X | X | |
| Muscle biopsy | | X | | | | | X | |
| Blood | | X | | X | | X | X | |
| U/S | | X | X | X | X | X | X | X |
| Functional | | | | | | | | X |
| testing | | | | | | | | |
| Balance Board | | | | | | | | X |
| Psychological | | | | | | | | X |

Heart monitoring and haemoglobin oxygen saturations will take place during cycling sessions.

Cycling will be daily, for 5 times per week.

## Appendix B - The CYCLE Trial Exclusion Criteria

## A. Daily exemption criteria for in-bed cycling

Cycling or physiotherapy (PT) sessions will not occur if any of the following conditions are present:

- 1. An increase in vasopressor/inotrope of more than 25% within past 2 h
- 2. Active myocardial ischaemia, or unstable/uncontrolled arrhythmia after discussion with the intensive care unit (ICU) team.
- 3. Mean arterial pressure (MAP) <60 or >110 mm Hg or out of range for this patient within the past 2 hours.
- 4. Heart rate <40 or >140 bpm within the past 2 hours.
- 5. Persistent SpO2 <88% or out of range for this patient within the past 2 hours.
- 6. Neuromuscular blocker within past 4 hours.
- 7. Severe agitation (Richmond Agitation and Sedation Scale >2 (or equivalent)) within past 2 hours.
- 8. Uncontrolled pain.
- 9. Change in goals to palliative care.
- 10. Team perception that in-bed cycling or therapy is not appropriate despite absence of above criteria (e.g., active major haemorrhage from any site, acute peritonitis, new incision or wound precluding cycling, new known/suspected muscle inflammation (e.g., rhabdomyolysis)).
- 11. Patient or proxy refusal.

## B. Criteria to terminate in-bed cycling or routine PT

Cycling or routine PT will stop if the following occurs:

- Concern for myocardial ischaemia or suspected new unstable/uncontrolled arrhythmia.
- 2. Unplanned extubation
- 3. Physiotherapist perceives continuing cycling or routine PT is not appropriate, for example,
- Respiratory—sustained O2 desaturation <88%; marked ventilator dysynchrony.
- Cardiovascular—sustained symptomatic bradycardia (<40 bpm), tachycardia (>140 bpm), hypotension (MAP <60 mm Hg) or hypertension (MAP >120 mm Hg).
- 6. Catheter or tube dislodgement or severe patient agitation.
- 7. ICU physician, patient or proxy requests termination of session.

## Appendix C - Proposed measurements and statistical test

An overview of all measurements and planned statistical analysis is presented in the table below. A p-value of less than 0.05 will be considered statistically significant.

## Appendix C - Proposed measurements and statistical test

An overview of all measurements and planned statistical analysis is presented in the table below. A p-value of less than 0.05 will be considered statistically significant.

Due to multiple comparisons, the Holm–Bonferroni method is used to control the group-wise error rate.

In all cases, a p-value of <0.05 after Holm–Bonferroni correction will be considered statistically significant.

| . w | I | | | | | | I |
|---|---|---|---|---|---|---|---|
| Category™ | Measurement | Units | Time@f@neasurement | Summary@Measure | Hypothesis@to@be@tested@HO-hypothesis) There@s@no@ifference@between@ntervention@ | Statistical@est | NOTES |
| Patienti Demographics | Age | Years | On@admission/consenting | Mean@ndlSD | and@ontrol@roup | UnpairedIt-test | |
| ratientabemographics | Age | rears | Ontadinission/consenting | | There@s@no@difference@between@ntervention@ | Onpaneda-test | |
| ' | Height | Metres | On@dmission/consenting | | and@ontrol@roup | Unpaired 1-test | |
| | | | | | Therellis@ho@difference@between@ntervention@ | | |
| | Weight | Kilograms | On@dmission/consenting | | and@tontrol@roup | Unpaired@-test | |
| | | | | | There@s@ho@difference@between@ntervention@ | | |
| | BMI | kg/m² | On@dmission/consenting | | anditontroligroup | Unpaired test | |
| <u>'</u> | | | | | There is thoughtference between intervention | | |
| | Sex | Count | On@admission/consenting | | | Chi-square@est | |
| <u>'</u> | APACHEDITScore | Arbitary@oints | On@admission/consenting | | Therelis Inold ifference Ibetween Intervention I and Itontroligroup | UnpairedIt-test | |
| | APACHEMISCORE | Arbitary#oints | Onladmission/consenting | MeanlandisD | andicontroligroup | Onpaireds-test | |
| | | | | | There@s@no@lifference@between@ntervention@ | | |
| (Vastusliateralis) | Musclethickness | Centimetres | Day[10] | Mean@hange@n@hickness@cm),@D | anditontroligroup | UnpairedII-test | |
| , | | | | | There@s@ho@difference@between@ntervention@ | | |
| | | | | Mean®@hange@n@hickness, &D | anditontroligroup | UnpairedIt-test | |
| | | | | Skew,@kurtosis | The data dare door mally distributed | Shapiro-Wilk | |
| | | | | | There@s@ho@difference@between@ntervention@ | | |
| Ultrasound | Fascicle@ennation@ngle | Degrees | Day11,13,15,17(1110,114 | Mean@hange@n@ngle@degrees), SD | anditontroligroup | Repeated measure analysis | |
| 1 | | | | | ThereIsinoldifferenceIbetweenIntervention | | |
| | | - | | | and@tontrol@roup | Repeated@neasure@analysis | |
| (Vastusliateralis,limediallimeadlibfili | Fasciclellength | Centimetres | Day(1,/3,/5,/7)(210,/14 | Mean@hange@n@ength@cm)@&D | There@s@no@ifference@between@ntervention@ | Repeated@neasure@analysis | |
| gastrochemius | rascicleidength | Cenumetres | Payid,id,id,id;id10,id4 | ivieanයnangeuniaengthii(cm)முக்ப | and@tontrol@roup There@s@ho@difference@between@ntervention@ | nepeateumeasure@naiysis | |
| 1 | | (Derived@byl@rigonometry) | | Mean®@thange@n@ength,@D | and@tontrol@roup | Repeated@neasure@nalvsis | FL=@hickness@Bin@Pennation@Angle) |
| | | (Sc., vediabyian gonometry) | | w.co.mouriangeanaengtii,abb | anazona ongroup | repeateumicasuretaridiysis | . z - w meknessyksmyr ennadonianigie) |
| | | | | | There@s@ho@difference@between@ntervention@ | | |
| Medial@head@f@astrocnemius | Muscle∄hickness | Centimetres | Day(1,13,15,17)(210,114 | Mean@thange@n@hickness@cm), SD | anditontroligroup | Repeated@neasure@nalysis | |
| | | | , | ,,_ | Therellis@holdifference@between@ntervention@ | | |
| <u>'</u> | | | | Mean Mathange In Thickness, SD | anditontroligroup | Repeated@neasure@nalysis | |
| | | | | | There is thoughtference between intervention | | |
| Rectus demoris, destus dateralis | Cross@ectional@rea | Square@entimetres | Day(1,13,15,17)(110,114 | Mean@hange@n@rea@cm²),[SD | anditontroligroup | Repeated@neasure@nalysis | |
| <u>'</u> | | | | | There@s@ho@difference@between@ntervention@ | | |
| Intermedius@nd@Medialis | | | | Mean Marea, SD | anditontroligroup | Repeated measure analysis | |
| la | | | | | Thereas a no difference between antervention | | |
| Rectus[Abdominis | Crossisectionaliarea | SquareCentimetres | Day(1,13,15,171)(10,114 | Meanlithangeliinläreali(cm²),ISD | and@tontrol@roup There@s@no@difference@between@ntervention@ | Repeatedlineasurellinalysis | |
| <u>'</u> | | | | Mean®©thange@nlarea,ISD | and@ontrol@roup | Repeatedlineasurellanalysis | |
| | | | | Weariowchangeunarea,iso | anditiontroligroup | Repeateumeasureamarysis | |
| | | | | | There is in ordifference between intervention | | |
| Diaphragm | Thickness | Centimetres | Day 11,13,15,17(1110,114 | Mean@thange@n@thickness@cm),@D | anditontroligroup | Repeated@measure@analysis | |
| - 1, | | | | | There is tho difference between intervention | , | |
| <u>'</u> | | | | Mean@@hange@n@hickness,@D | and@tontroll@roup | Repeated@neasure@analysis | |
| | | | | - | There is in ordifference between intervention | | |
| All@nuscles | Echogenicity | Arbitary, Scale from 10-1 | Day[1,/10. | Change In Echogenicity, ISD | anditontroligroup | UnpairedIt-test | |
| <u>'</u> | | | | | ThereIIsIholdifferenceIbetweenIIntervention | | |
| Diaphragm | Thickening: Fraction | Percentage | Day/1,/3,/5,/7/2/10,/14 | Mean@thange@n@Fraction@(%)@D | andlitontrolligroup | Logiliankiitest | |
| l ' | | | | | Therelistholdifferencelbetweenlintervention | | |
| Diaphragm | MaximalExcursion | Centimetres | Day(1,8,5,7)(10,14 | Mean@hange@n@xcursion@cm),&D | anditontroligroup | Log@ank@est | |
| <u> </u> | | - | | | There@s@no@torrelation@between@muscle@ | | |
| 1 | Change@n@nuscle@hickness@n@day@ | | | | thickness@n@dav@10@nd@ | | |
| 1 | 10@elated@o@ge/weight/baseline@ | | | | age/weight/baseline@muscle@hickness@ | | |
| Measures@f@orrelation | | Centimetres@s@rs/kg/cm | Losses@by@day@10 | | betwen@ntervention@nd@ontrol@roup | Pearson's test | |
| | 1 | 7.77.00 | | | | | |
| Biochemical desting | | | | | | | |
| MuscleBiopsy | | TBC | | | | TBC | |
| Blood/Urine | TBC | TBC | Day@1,65,67,@10 | TBC | ТВС | TBC | |
| Follow@up@measures | | | | | | | |
| Dynamometry | Handigrip | Newtons | | Mean@ifference@n@orce@N), ISD. | | unpaired@t-test | |
| Dynamometry | | Newtons | | Mean@difference@n@force@N), (SD. | | unpaired t-test | |
| 6@ninute@walk@est | | Metres | | Mean@ifference@n@istance@metres),(\$D | | unpaired 1-test | |
| Ultrasoundiīvastusilateralis | | Centremeters | | Mean@ifference@n@hickness@cm),(SD | | unpaired@test | |
| SF-36/3core<br>Balance | | Arbitary@oints | At@months#/U@ppointment | | | unpaired@test | |
| Balance<br>MRClSumiPowerlScore | Average\(\mathbb{S}\)way Total\(\mathbb{S}\)core | Arbitary@from@-36@oints | Ati3@monthsi#/U@ppointment Ati3@monthsi#/U@ppointment | | | unpairedIt-test | |
| | rotalipeore | Arbitarymanoritus-souponits | Account is any orappoint ment | wearium erenceuriscore,iso | | unpan cuta-test | |
| on Page | | | | | | | |
| Incidence of delirium | Count | Count@nd® | From@ays@1-14 | Perecentage@ifference | | Chi-squaretestatisher's@xacttest | |
| Incidence@fileeding@RRT | | Count@nd@6 | | Perecentage@difference | | Chi-squarellest@fisher's@xactilest | |
| Safety@tubes/lines@ulled | | Count@nd@ | From@days@1-14 | Perecentage difference | | Chi-squarellest@fisher's@xactllest | |
| | | - | | | | | |

- 1. Kizilarslanoglu MC, Kuyumcu ME, Yesil Y, Halil M. Sarcopenia in critically ill patients. J Anesth [Internet]. 2016 Oct 4 [cited 2018 Apr 9];30(5):884–90. Available from: http://link.springer.com/10.1007/s00540-016-2211-4
- 2. Stevens RD, Marshall SA, Cornblath DR, Hoke A, Needham DM, de Jonghe B, et al. A framework for diagnosing and classifying intensive care unit-acquired weakness. Crit Care Med [Internet]. 2009 Oct [cited 2018 Apr 9];37(10 Suppl):S299–308. Available from: http://www.ncbi.nlm.nih.gov/pubmed/20046114
- 3. Herridge MS, Tansey CM, Matté A, Tomlinson G, Diaz-Granados N, Cooper A, et al. Functional Disability 5 Years after Acute Respiratory Distress Syndrome. N Engl J Med [Internet]. 2011 Apr 7 [cited 2018 Apr 9];364(14):1293–304. Available from: http://www.nejm.org/doi/abs/10.1056/NEJMoa1011802
- 4. Yende S, Austin S, Rhodes A, Finfer S, Opal S, Thompson T, et al. Long-Term Quality of Life Among Survivors of Severe Sepsis: Analyses of Two International Trials. Crit Care Med [Internet]. 2016 Aug [cited 2018 Apr 9];44(8):1461–7. Available from: http://www.ncbi.nlm.nih.gov/pubmed/26992066
- 5. Kress J, Herridge M. Medical and Economic Implications of Physical Disability of Survivorship. Semin Respir Crit Care Med [Internet]. 2012 Aug 8 [cited 2018 Apr 9];33(4):339–47. Available from: http://www.ncbi.nlm.nih.gov/pubmed/22875379
- 6. Parry SM, El-Ansary D, Cartwright MS, Sarwal A, Berney S, Koopman R, et al. Ultrasonography in the intensive care setting can be used to detect changes in the quality and quantity of muscle and is related to muscle strength and function. J Crit Care [Internet]. 2015 Oct [cited 2018 Apr 9];30(5):1151.e9-1151.e14. Available from: http://www.ncbi.nlm.nih.gov/pubmed/26211979
- 7. Turton P, Hay R, Taylor J, McPhee J, Welters I. Human limb skeletal muscle wasting and architectural remodeling during five

- to ten days intubation and ventilation in critical care an observational study using ultrasound. BMC Anesthesiol [Internet]. 2016 [cited 2018 Mar 18];16(1):119. Available from: http://www.ncbi.nlm.nih.gov/pubmed/27894277
- 8. Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, et al. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med [Internet]. 2013 May 24 [cited 2018 Apr 9];39(5):801–10. Available from: http://www.ncbi.nlm.nih.gov/pubmed/23344830
- 9. Walker FO, Cartwright MS, Wiesler ER, Caress J. Ultrasound of nerve and muscle. Clin Neurophysiol [Internet]. 2004 Mar 1 [cited 2018 Apr 9];115(3):495–507. Available from: http://www.ncbi.nlm.nih.gov/pubmed/15036045
- 10. Fivez T, Hendrickx A, Van Herpe T, Vlasselaers D, Desmet L, Van den Berghe G, et al. An Analysis of Reliability and Accuracy of Muscle Thickness Ultrasonography in Critically III Children and Adults. J Parenter Enter Nutr [Internet]. 2016 Sep 11 [cited 2018 Apr 9];40(7):944–9. Available from: http://doi.wiley.com/10.1177/0148607115575033
- de Boer MD, Seynnes OR, di Prampero PE, Pišot R, Mekjavić IB, Biolo G, et al. Effect of 5 weeks horizontal bed rest on human muscle thickness and architecture of weight bearing and non-weight bearing muscles. Eur J Appl Physiol [Internet].
   2008 Sep 5 [cited 2018 Apr 9];104(2):401–7. Available from: http://www.ncbi.nlm.nih.gov/pubmed/18320207
- 12. Gruther W, Benesch T, Zorn C, Paternostro-Sluga T, Quittan M, Fialka-Moser V, et al. Muscle wasting in intensive care patients: Ultrasound observation of the M. quadriceps femoris muscle layer. J Rehabil Med [Internet]. 2008 Mar [cited 2018 Apr 2];40(3):185–9. Available from: http://www.ncbi.nlm.nih.gov/pubmed/18292919
- 13. Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, et al. Acute Skeletal Muscle Wasting in Critical Illness. JAMA [Internet]. 2013 Oct 16 [cited 2018 Apr 2];310(15):1591. Available from: http://www.ncbi.nlm.nih.gov/pubmed/24108501

- 14. Calvo-Ayala E, Khan BA, Farber MO, Ely EW, Boustani MA. Interventions to improve the physical function of ICU survivors: a systematic review. Chest [Internet]. 2013 Nov [cited 2018 Apr 9];144(5):1469–80. Available from: http://www.ncbi.nlm.nih.gov/pubmed/23949645
- 15. Kho ME, Molloy AJ, Clarke F, Herridge MS, Koo KKY, Rudkowski J, et al. CYCLE pilot: a protocol for a pilot randomised study of early cycle ergometry versus routine physiotherapy in mechanically ventilated patients. BMJ Open [Internet]. 2016 Apr 8 [cited 2018 Apr 9];6(4):e011659. Available from: http://www.ncbi.nlm.nih.gov/pubmed/27059469
- 16. Camargo Pires-Neto R, Fogaça Kawaguchi YM, Sayuri Hirota A, Fu C, Tanaka C, Caruso P, et al. Very Early Passive Cycling Exercise in Mechanically Ventilated Critically III Patients: Physiological and Safety Aspects A Case Series. Lucia A, editor. PLoS One [Internet]. 2013 Sep 9 [cited 2018 Apr 9];8(9):e74182. Available from: http://dx.plos.org/10.1371/journal.pone.0074182
- 17. dos Santos LJ, de Aguiar Lemos F, Bianchi T, Sachetti A, Dall' Acqua AM, da Silva Naue W, et al. Early rehabilitation using a passive cycle ergometer on muscle morphology in mechanically ventilated critically ill patients in the Intensive Care Unit (MoVe-ICU study): study protocol for a randomized controlled trial. Trials [Internet]. 2015 Aug 28 [cited 2018 Apr 9];16:383. Available from: http://www.ncbi.nlm.nih.gov/pubmed/26314881
- 18. Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, et al. Early exercise in critically ill patients enhances short-term functional recovery\*. Crit Care Med [Internet]. 2009 Sep [cited 2018 Apr 9];37(9):2499–505. Available from: http://www.ncbi.nlm.nih.gov/pubmed/19623052
- 19. Lee D, Lee G, Jeong J. Mirror Therapy with Neuromuscular Electrical Stimulation for improving motor function of stroke survivors: A pilot randomized clinical study. Technol Heal Care [Internet]. 2016 Jul 27 [cited 2018 Apr 9];24(4):503–11. Available from: http://www.ncbi.nlm.nih.gov/pubmed/26890230

- 20. Fischer A, Spiegl M, Altmann K, Winkler A, Salamon A, Themessl-Huber M, et al. Muscle mass, strength and functional outcomes in critically ill patients after cardiothoracic surgery: does neuromuscular electrical stimulation help? The Catastim 2 randomized controlled trial. Crit Care [Internet]. 2016 Dec 29 [cited 2018 Apr 9];20(1):30. Available from: http://www.ncbi.nlm.nih.gov/pubmed/26825278
- 21. Kho ME, Truong AD, Zanni JM, Ciesla ND, Brower RG, Palmer JB, et al. Neuromuscular electrical stimulation in mechanically ventilated patients: A randomized, sham-controlled pilot trial with blinded outcome assessment. J Crit Care [Internet]. 2015 Feb [cited 2018 Apr 9];30(1):32–9. Available from: http://www.ncbi.nlm.nih.gov/pubmed/25307979
- 22. Segers J, Hermans G, Bruyninckx F, Meyfroidt G, Langer D, Gosselink R. Feasibility of neuromuscular electrical stimulation in critically ill patients. J Crit Care [Internet]. 2014 Dec [cited 2018 Apr 9];29(6):1082–8. Available from: http://www.ncbi.nlm.nih.gov/pubmed/25108833
- 23. Bauer P, Krewer C, Golaszewski S, Koenig E, Müller F. Functional Electrical Stimulation—Assisted Active Cycling—
  Therapeutic Effects in Patients With Hemiparesis From 7 Days to 6 Months After Stroke: A Randomized Controlled Pilot Study. Arch Phys Med Rehabil [Internet]. 2015 Feb [cited 2018 Apr 9];96(2):188–96. Available from:
  http://www.ncbi.nlm.nih.gov/pubmed/25449195
- 24. Ambrosini E, Ferrante S, Pedrocchi A, Ferrigno G, Molteni F. Cycling Induced by Electrical Stimulation Improves Motor Recovery in Postacute Hemiparetic Patients: A Randomized Controlled Trial. Stroke [Internet]. 2011 Apr 1 [cited 2018 Apr 9];42(4):1068–73. Available from: http://www.ncbi.nlm.nih.gov/pubmed/21372309
- 25. Lo H-C, Hsu Y-C, Hsueh Y-H, Yeh C-Y. Cycling exercise with functional electrical stimulation improves postural control in stroke patients. Gait Posture [Internet]. 2012 Mar [cited 2018 Apr 9];35(3):506–10. Available from: http://www.ncbi.nlm.nih.gov/pubmed/22153770

- 26. Parry SM, Berney S, Warrillow S, El-Ansary D, Bryant AL, Hart N, et al. Functional electrical stimulation with cycling in the critically ill: A pilot case-matched control study. J Crit Care [Internet]. 2014 Aug [cited 2018 Apr 9];29(4):695.e1-695.e7. Available from: http://www.ncbi.nlm.nih.gov/pubmed/24768534
- 27. Needham DM, Truong AD, Fan E. Technology to enhance physical rehabilitation of critically ill patients. Crit Care Med [Internet]. 2009 Oct [cited 2018 Apr 9];37(10 Suppl):S436–41. Available from: http://www.ncbi.nlm.nih.gov/pubmed/20046132
- 28. Parry SM, Berney S, Koopman R, Bryant A, El-Ansary D, Puthucheary Z, et al. Early rehabilitation in critical care (eRiCC): functional electrical stimulation with cycling protocol for a randomised controlled trial. BMJ Open [Internet]. 2012 Jan 1 [cited 2018 Apr 9];2(5):e001891. Available from: http://www.ncbi.nlm.nih.gov/pubmed/22983782
- 29. Kandarian SC, Jackman RW. Intracellular signaling during skeletal muscle atrophy. Muscle Nerve [Internet]. 2006 Feb [cited 2018 Apr 9];33(2):155–65. Available from: http://www.ncbi.nlm.nih.gov/pubmed/16228971
- 30. Eikermann M, Koch G, Gerwig M, Ochterbeck C, Beiderlinden M, Koeppen S, et al. Muscle force and fatigue in patients with sepsis and multiorgan failure. Intensive Care Med [Internet]. 2006 Feb 27 [cited 2018 Apr 9];32(2):251–9. Available from: http://www.ncbi.nlm.nih.gov/pubmed/16468072
- 31. Jackman RW, Cornwell EW, Wu C-L, Kandarian SC. Nuclear factor-κB signalling and transcriptional regulation in skeletal muscle atrophy. Exp Physiol [Internet]. 2013 Jan [cited 2018 Apr 9];98(1):19–24. Available from: http://www.ncbi.nlm.nih.gov/pubmed/22848079
- 32. Ho RC, Hirshman MF, Li Y, Cai D, Farmer JR, Aschenbach WG, et al. Regulation of IκB kinase and NF-κB in contracting adult rat skeletal muscle. Am J Physiol Physiol [Internet]. 2005 Oct [cited 2018 Apr 9];289(4):C794–801. Available from: http://www.ncbi.nlm.nih.gov/pubmed/15888549

- 33. KUMAR A, BORIEK AM. Mechanical stress activates the nuclear factor-kappaB pathway in skeletal muscle fibers: a possible role in Duchenne muscular dystrophy. FASEB J [Internet]. 2003 Mar [cited 2018 Apr 9];17(3):386–96. Available from: http://www.ncbi.nlm.nih.gov/pubmed/12631578
- 34. JI LL, GOMEZ-CABRERA M-C, STEINHAFEL N, VINA J. Acute exercise activates nuclear factor (NF)-κB signaling pathway in rat skeletal muscle. FASEB J [Internet]. 2004 Oct [cited 2018 Apr 9];18(13):1499–506. Available from: http://www.ncbi.nlm.nih.gov/pubmed/15466358
- 35. McGlory C, Phillips SM. Assessing the regulation of skeletal muscle plasticity in response to protein ingestion and resistance exercise. Curr Opin Clin Nutr Metab Care [Internet]. 2014 Sep [cited 2018 Apr 9];17(5):412–7. Available from: http://www.ncbi.nlm.nih.gov/pubmed/25105927
- 36. Jackson MJ, McArdle A. Age-related changes in skeletal muscle reactive oxygen species generation and adaptive responses to reactive oxygen species. J Physiol [Internet]. 2011 May 1 [cited 2018 Apr 9];589(9):2139–45. Available from: http://www.ncbi.nlm.nih.gov/pubmed/21320885
- 37. Pedersen BK, Febbraio MA. Muscles, exercise and obesity: skeletal muscle as a secretory organ. Nat Rev Endocrinol [Internet]. 2012 Aug 3 [cited 2018 Apr 9];8(8):457–65. Available from: http://www.ncbi.nlm.nih.gov/pubmed/22473333
- 38. Witteveen E, Wieske L, van der Poll T, van der Schaaf M, van Schaik IN, Schultz MJ, et al. Increased Early Systemic Inflammation in ICU-Acquired Weakness; A Prospective Observational Cohort Study\*. Crit Care Med [Internet]. 2017 Jun [cited 2018 Apr 9];45(6):972–9. Available from: http://www.ncbi.nlm.nih.gov/pubmed/28350642
- 39. Bolton CF. Neuromuscular manifestations of critical illness. Muscle Nerve [Internet]. 2005 Aug 1 [cited 2018 Apr 9];32(2):140–63. Available from: http://doi.wiley.com/10.1002/mus.20304

- 40. Jones S, Chiesa ST, Chaturvedi N, Hughes AD. Recent developments in near-infrared spectroscopy (NIRS) for the assessment of local skeletal muscle microvascular function and capacity to utilise oxygen. Artery Res [Internet]. 2016 Dec [cited 2018 Apr 9];16:25–33. Available from: http://www.ncbi.nlm.nih.gov/pubmed/27942271
- 41. Maffiuletti NA, Roig M, Karatzanos E, Nanas S. Neuromuscular electrical stimulation for preventing skeletal-muscle weakness and wasting in critically ill patients: a systematic review. [cited 2018 Apr 9]; Available from: https://bmcmedicine.biomedcentral.com/track/pdf/10.1186/1741-7015-11-137
- 42. Acqua A, Sachetti A, Santos L, Lemos F, Bianchi T, Naue W, et al. Use of neuromuscular electrical stimulation to preserve the thickness of abdominal and chest muscles of critically ill patients: A randomized clinical trial. J Rehabil Med [Internet]. 2017 Jan 19 [cited 2018 Apr 9];49(1):40–8. Available from: http://www.ncbi.nlm.nih.gov/pubmed/28101565
- 43. Cho HK, Jung GS, Kim EH, Cho YW, Kim SW, Ahn SH. The effects of neuromuscular electrical stimulation at different frequencies on the activations of deep abdominal stabilizing muscles. J Back Musculoskelet Rehabil [Internet]. 2016 Jan 25 [cited 2018 Apr 9];29(1):183–9. Available from: http://www.ncbi.nlm.nih.gov/pubmed/26444328
- 44. Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, et al. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA [Internet]. 2016 Feb 23 [cited 2018 Apr 9];315(8):801. Available from: http://jama.jamanetwork.com/article.aspx?doi=10.1001/jama.2016.0287
- 45. Nakanishi N, Oto J, Tsutsumi R, Iuchi M, Onodera M, Nishimura M. Upper and lower limb muscle atrophy in critically ill patients: an observational ultrasonography study. Intensive Care Med [Internet]. 2018 Feb [cited 2018 Mar 18];44(2):263–4. Available from: http://www.ncbi.nlm.nih.gov/pubmed/29110031
- 46. Shanely RA, Zwetsloot KA, Triplett NT, Meaney MP, Farris GE, Nieman DC. Human Skeletal Muscle Biopsy Procedures

Using the Modified Bergström Technique. J Vis Exp [Internet]. 2014 Sep 10 [cited 2018 Apr 9];(91):51812. Available from: http://www.ncbi.nlm.nih.gov/pubmed/25285722

47. Bergstrom J. Percutaneous needle biopsy of skeletal muscle in physiological and clinical research. Scand J Clin Lab Invest [Internet]. 1975 Nov [cited 2018 Apr 9];35(7):609–16. Available from: http://www.ncbi.nlm.nih.gov/pubmed/1108172